CLINICAL TRIAL: NCT02925195
Title: Multi Ethnic Study of Atherosclerosis Individualized Response to Vitamin D Treatment Study
Brief Title: Individualized Response to Vitamin D Treatment Study
Acronym: INVITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ian deBoer, Associate Professor, Medicine/Nephrology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001485; R01HL096875 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Characteristics That Modify the Response to Cholecalciferol Treatment
Keywords: Vitamin D; cardiovascular disease; MESA; genetics; pharmacogenetics; blood pressure; biomarkers
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — cholecalciferol (vitamin D3) 2000 IU capsules daily
  Arms: Active Treatment
Drug: Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine individual-level genetic and metabolic characteristics that modify the response to cholecalciferol treatment.

This study is double blind, parallel design, randomized clinical trial that will assess genetic and metabolic characteristics that modify the response to cholecalciferol treatment. . Eligible participants will be randomly assigned to receive cholecalciferol treatment (2,000 international units of cholecalciferol daily by mouth) or placebo in a 3:1 ratio for a total duration of 16-weeks. The planned sample size is 1,600. The primary aim of this study is to identify genetic polymorphisms, clinical characteristics, and biomarkers that modify the biologic response to vitamin D3 treatment, assessed by changes in serum concentrations of parathyroid hormone (PTH) and 1,25(OH)2D and urine calcium excretion.

ELIGIBILITY:
Inclusion Criteria:

1,600 participants from the Multi-Ethnic Study of Atherosclerosis (MESA) study who are returning for their scheduled 6th MESA study visit.

Participants will be recruited from four field centers: Wake Forest University, Winston-Salem, NC; Columbia University, New York, NY; Northwestern University, Evanston, IL; and Johns Hopkins University, Baltimore, MD.

Exclusion Criteria:

1. Current use of >1,000 international units (IU) of cholecalciferol daily
2. Current use of any activated vitamin D product (calcitriol, paricalcitol, hectorol)
3. Known history of allergy or adverse reaction to vitamin D treatment
4. Known clinical history of primary hyperparathyroidism
5. Known clinical history of kidney stones within the previous 5 years
6. Current participation in another interventional study
7. Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, Principal Investigator — University of Washington; Bryan Kestenbaum, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Northwestern University, Evanston, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Columbia Univeristy, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Hsu S, Prince DK, Williams K, Allen NB, Burke GL, Hoofnagle AN, Li X, Liu KJ, McClelland RL, Michos ED, Psaty BM, Shea SJ, Rice KM, Rotter JI, Siscovick D, Tracy RP, Watson KE, Kestenbaum BR, de Boer IH. Clinical and biomarker modifiers of vitamin D treatment response: the Multi-Ethnic Study of Atherosclerosis. Am J Clin Nutr. 2022 Mar 4;115(3):914-924. doi: 10.1093/ajcn/nqab390. PMID 34849546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 499 | 167
Completed | 453 | 158
Not Completed | 46 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 499 | 167 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8) | 72 (8) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 81 | 353
  Male | 227 | 86 | 313
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 169 | 58 | 227
  Non-Hispanic Black | 184 | 61 | 245
  Chinese | 64 | 19 | 83
  Hispanic | 82 | 29 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum 1,25(OH)2D Concentration
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 499 | 167
pg/mL | 2 (16) | -1 (17)

2. Primary Outcome: Change in Serum PTH Concentration
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 499 | 167
pg/mL | -3 (16) | 2 (18)

3. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 499 | 167
mmHg | -3 (18) | -4 (16)

4. Secondary Outcome: Change in Urine Calcium Excretion
Description: Urine calcium excretion estimated as spot urine calcium-creatinine ratio
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mg per g of creatinine
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 499 | 167
mg per g of creatinine | 8 (83) | 1 (70)

5. Secondary Outcome: Change in Serum Calcium Concentrations
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 499 | 167
mg/dL | 0 (0.3) | 0 (0.3)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Active Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 1/499 | 0/167
Serious Adverse Events (participants affected / at risk) | 2/499 | 2/167
Other Adverse Events (participants affected / at risk) | 55/499 | 16/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=499) | Placebo (N=167)
Diverticulosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=499) | Placebo (N=167)
Cardiac disorders (Cardiac disorders) | 5 (5) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 22 (22) | 6 (6)
General disorders and administration site conditions (General disorders) | 8 (8) | 1 (1)
Immune system disorders (Immune system disorders) | 8 (8) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Musculoskeletal, connective tissue, and bone disorders (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary tract disorders (Renal and urinary disorders) | 1 (1) | 2 (2)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
(General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02925195/Prot_SAP_000.pdf